CLINICAL TRIAL: NCT07121569
Title: Efficacy of Oral DLBS1033 as Adjunctive Therapy in Acute Ischemic Stroke: A Randomized Controlled Trial Evaluating Inflammatory Biomarkers, TCD Results, and Clinical Outcomes
Brief Title: Oral DLBS1033 as Adjunctive Therapy in Acute Ischemic Stroke: Impact on Inflammatory Biomarkers and Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Firstiafina Tiffany, Medical Doctor (Neurologist), Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLBS1033 on Ischemic Stroke; UST-003.24/DLBS1033/1/2024 (Other: Grantor or Funder: Dexa Medica Group)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke, Acute
Keywords: Interleukin-6; Ischemic Stroke; Treatment outcome; Tumor Necrosis Factor-alpha; Oral lumbrokinase DLBS1033
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This randomized, double-masked controlled trial employed a rigorous experimental design to compare the adjunctive therapeutic effects of oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica, 2 tab t.i.d.) versus placebo in patients with acute ischemic stroke over a 28-day prospective observation period. The study was conducted in the inpatient ward, with follow-up at the outpatient clinic of the Neurology Department, Dr. Moewardi General Hospital, Surakarta, Central Java, Indonesia, from July 2024 to March 2025, after obtaining full ethical clearance from the hospital's Health Research Ethics Committee
Who Masked: Participant, Investigator
Masking Description: The study utilized a two-block randomization method to achieve balanced group assignments. Random allocation sequences were prepared by independent personnel and secured in sealed envelope. Each treatment package was labeled with a subject identification number corresponding to the generated random sequence and was distributed to eligible participants. The codes were kept confidential until the study was completed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral lumbrokinase DLBS1033 group (Experimental): Patients with acute ischemic stroke who received oral lumbrokinase DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica, 2 tabs t.i.d.) and 100 mg acetylsalicylic acid as standard stroke therapy during 28-days observation period
  Interventions: Drug: Oral lumbrokinase DLBS1033
- Placebo group (Active Comparator): Patients with acute ischemic stroke who received placebo (Placebo by Dexa Medica, 2 tabs t.i.d.) and 100 mg acetylsalicylic acid as standard stroke therapy during 28-days observation period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral lumbrokinase DLBS1033 — DLBS1033: 490 mg, DISOLF film-coated tablet, Dexa Medica, 2 tabs t.i.d
  Other Names: DISOLF
  Arms: Oral lumbrokinase DLBS1033 group
Drug: Placebo — Placebo by Dexa Medica, 2 tabs t.i.d.
  Arms: Placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled trial aims to evaluate the effect of oral DLBS1033 as adjunctive therapy on inflammatory biomarkers (IL-6, TNF-α, MMP-9, D-dimer), transcranial Doppler (TCD) parameters, and clinical outcomes in patients with acute ischemic stroke. Fifty-two eligible patients admitted to RSUD Dr. Moewardi Surakarta will be randomly assigned to receive either DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica, 2 tab t.i.d.) or placebo for 28 days, in addition to standard therapy between July 2024 to March 2025. The study was conducted in the inpatient ward, with follow-up at the outpatient clinic of the Neurology Department, Dr. Moewardi General Hospital, Surakarta, Central Java, following full ethical approval from the hospital's Health Research Ethics Committee. Primary outcomes include changes in inflammatory markers; secondary outcomes include changes in NIHSS and Barthel Index scores and TCD profiles.

DETAILED DESCRIPTION:
Intravenous thrombolysis with tissue plasminogen activator (tPA) or mechanical thrombectomy is considered first-line treatment to mediate reperfusion. Despite the rapid restoration of cerebral blood flow post-stroke, recanalization of occluded vessels can lead to progressive tissue damage, a condition known as ischemia-reperfusion injury. Reperfusion triggers a strong inflammatory response, supporting the development of a thrombo-inflammatory cascade. Previous studies have shown that lumbrokinase, a component of DLBS1033, plays a role in modulating the inflammatory cascade. Lumbrokinase has been shown to significantly reduce several inflammatory biomarkers, such as IL-6, TNF-alpha, and MMP-9, in an animal study level. However, no studies have yet examined the role of lumbrokinase in reducing TNF-α, MMP-9, and IL-6 levels in the blood of patients with ischemic stroke. Previous studies stated that administration of DLBS1033 significantly improves clinical outcomes in ischemic stroke patients, as measured by NIHSS and Barthel Index scores. Based on this background, the researcher is interested in investigating the effect of oral DLBS1033 as adjunctive therapy on the thrombo-inflammatory patho-mechanism in patients with ischemic stroke, as assessed by inflammatory biomarkers, TCD parameters, and clinical outcomes.

Eligible patients diagnosed with acute ischemic stroke, presenting within a time window of 24 hours to 7 days from symptom onset, will be enrolled and randomly assigned into two parallel groups in a 1:1 ratio. The diagnosis of ischemic stroke was made based on physical examination and confirmed by a non-contrast head CT scan performed by a neurologist. One group will receive oral DLBS1033 (490 mg, DISOLF film-coated tablet, Dexa Medica, 2 tab t.i.d.), while the other will receive a matching placebo. Both interventions will be administered alongside standard stroke treatment protocols for a duration of 28 days. Randomization will be stratified to ensure balanced baseline characteristics between groups. Random allocation sequences were prepared by independent team and secured in sealed envelope. Each treatment package was pre-labeled with a unique subject identification number that corresponded to the assigned number in the randomization sequence. Upon enrollment, eligible participants received the treatment package that matched their assigned number.

Throughout the study, several key parameters will be assessed to evaluate the efficacy and safety of DLBS1033 as an adjunctive therapy. These include inflammatory biomarkers, such as serum levels of interleukin-6 (IL-6), tumor necrosis factor-alpha (TNF-α), matrix metalloproteinase-9 (MMP-9), and D-dimer, which will be measured using validated immunoassay methods. In addition, cerebral hemodynamic status will be evaluated through Transcranial Doppler (TCD) ultrasonography to assess Pulsatility Index (PI), and carotid intima-media thickness (CIMT) will be measured via B-mode ultrasonography to examine vascular structural changes.

To evaluate clinical outcomes, the National Institutes of Health Stroke Scale (NIHSS) will be used to assess neurological deficits, and the Barthel Index will be used to evaluate functional independence in daily activities. All assessments, including laboratory biomarker tests, TCD and CIMT measurements, and clinical outcome scoring, will be conducted at three key time points: baseline, day 14, and day 28 post-initiation of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient with acute ischemic stroke onset 24 hours-7 days confirmed by CT scan.
* First-ever or recurrent ischemic stroke.
* Compos mentis on admission.
* NIHSS score 5-25 on admission.
* Willing to participate and signed informed consent

Exclusion Criteria:

* Hemorrhagic stroke within the last 3 months.
* Transient ischemic attack.
* Pregnant, breastfeeding, or planning pregnancy.
* Use of anticoagulants in the past month.
* Nasogastric tube feeding.
* Having or History of bleeding disorders or coagulopathy.
* History of autoimmune disease.
* Severe renal impairment (serum creatinine ≥3× normal or on hemodialysis).
* Acute infection (systemic inflammatory response syndrome).
* Hypersensitivity to DLBS1033

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-07-06 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
MMP-9 | Baseline, day 14 and 28
  The inflammatory biomarkers were measured on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28
IL-6 | Baseline, day 14 and 28
  The inflammatory biomarkers were measured on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28
TNF-alpha | Baseline, day 14 and 28
  The inflammatory biomarkers were measured on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28
d-dimer | Baseline, day 14 and 28
  The inflammatory biomarkers were measured on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28

SECONDARY OUTCOMES:
TCD parameter-CIMT | Baseline, day 14 and 28
  Measurement of carotid intima-media thickness using TCD examination of the CCA was performed on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28. CIMT values fall within a positive range, greater than 0, where higher values indicate a possible thickening of the blood vessels, as a sign of atherosclerosis
TCD parameter-PI | Baseline, day 14 and 28
  Measurement of the pulsatility index using TCD examination of the CCA, ICA, vertebral artery, MCA, ACA, PCA, and ROA was conducted on the day of admission for stroke onset of 4-7 days, or on the third day for stroke onset of 1-3 days, and after the patient had received therapy on days 14 and 28. PI values fall within a positive range, greater than 0, where higher values indicate greater vascular resistance.
NIHSS | Baseline, day 14 and 28
  Assessment of stroke severity was conducted by evaluating various neurological functions, including consciousness, gaze, visual field, facial palsy, extrimity function, ataxia, sensory, language, dysarthria, and aphasia. This assessment was performed before the patient received therapy and after the patient had undergone therapy for 14 and 28 days. Minimum score is 0 and maximum score is 42, where a higher NIHSS score indicates a more severe degree of stroke.
Barthel Index | Baseline, day 14 and 28
  Assessment of the ability to perform activities of daily living, such as eating, drinking, self-care, mobility, using the toilet, moving around, climbing stairs, dressing, and bladder and bowel control, was conducted before the patient received therapy and after the patient had undergone therapy for 14 and 28 days. Minimum score is 0 and maximum score is 100, where a higher Barthel Index score indicates better patient ADL function.

CONTACTS AND LOCATIONS:
Overall Officials: Firstiafina Tiffany, MD, Principal Investigator — Department of Neurology, Faculty of Medicine, Universitas Sebelas Maret
Locations (1):
- Dr. Moewardi Regional General Hospital, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Publication in ICMJE journals
Supporting Information: Study Protocol, SAP, CSR
Time Frame: August 6th, 2025-August 6th, 2026
Access Criteria: Open access, every journal visitor

REFERENCES:
- [Background] Pinzon RT, Tjandrawinata RR, Wijaya VO, Veronica V. Effect of DLBS1033 on Functional Outcomes for Patients with Acute Ischemic Stroke: A Randomized Controlled Trial. Stroke Res Treat. 2021 Apr 7;2021:5541616. doi: 10.1155/2021/5541616. eCollection 2021. PMID 33927846
- [Background] Wang WL, Hsu YM, Lin ML, Chen SS, Lai YH, Huang CH, Yao CH. Ex Vivo Model to Evaluate the Antibacterial and Anti-Inflammatory Effects of Gelatin-Tricalcium Phosphate Composite Incorporated with Emodin and Lumbrokinase for Bone Regeneration. Bioengineering (Basel). 2023 Jul 31;10(8):906. doi: 10.3390/bioengineering10080906. PMID 37627791
- See also: Related Info — https://perpustakaan.rsmoewardi.com/index.php?p=show_detail&id=1645&keywords=Dlbs1033